CLINICAL TRIAL: NCT00661895
Title: Black Education and Treatment of Hypertension (BEAT HTN)
Acronym: BEAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-13859; 05-13589 (Other: Creighton University Institutional Review Board)
Record Dates: First submitted 2007-12-28; First posted 2008-04-21 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Hypertension
Keywords: African American
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Lisinopril; hydrochlorothiazide, lisinopril drug combination; Nifedipine; Metoprolol; Atenolol; Valsartan; Doxazosin; Clonidine; Hydralazine; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention group subjects will receive education and assistance from a Community Health Center or Cardiac Center nurse practitioner or physician, health educator, dietitian, social worker, and Cardiac Center-trained community members called Community Health Advocates (CHAs).
  Interventions: Drug: Hydrochlorothiazide; Drug: Lisinopril; Drug: Lisinopril and Hydrochlorothiazide; Drug: Nifedipine XL; Drug: Metoprolol tartrate; Drug: Atenolol; Drug: Valsartan; Drug: Doxazosin; Drug: Clonidine; Drug: Hydralazine; Drug: Metoprolol succinate; Drug: Amlodipine
- Control (Active Comparator): No intervention
  Interventions: Drug: Hydrochlorothiazide; Drug: Lisinopril; Drug: Lisinopril and Hydrochlorothiazide; Drug: Nifedipine XL; Drug: Metoprolol tartrate; Drug: Atenolol; Drug: Valsartan; Drug: Doxazosin; Drug: Clonidine; Drug: Hydralazine; Drug: Metoprolol succinate; Drug: Amlodipine

INTERVENTIONS:
Drug: Hydrochlorothiazide — Hydrochlorothiazide 25 mg tablets
Drug: Lisinopril — Lisinopril 5mg Tablet, 10 mg tablet, 20 mg tablet
Drug: Lisinopril and Hydrochlorothiazide — L 10 mg and H 12.5 mg tablets, L 20 mg and H 12.5 mg tablets, L 20 mg and H 25 mg tablets
Drug: Nifedipine XL — 30 mg extended release tablets, 60 mg extended release tablets
Drug: Metoprolol tartrate — 50 mg tablets & 100 mg tablets
  Other Names: Lopressor
Drug: Atenolol — 50 mg tablet
Drug: Valsartan — 80 mg tablets & 160 mg tablet
Drug: Doxazosin — 4 mg tablets
Drug: Clonidine — 0.2 mg tablets
Drug: Hydralazine — 50 mg tablets
Drug: Metoprolol succinate — 50 mg tablet & 100 mg tablet
  Other Names: Toprol XL
Drug: Amlodipine — 5 mg tablets & 10 mg tablets
  Other Names: Norvasc

SUMMARY:
Clinical trials have yet to test the adequacy of HTN control in African Americans (AA) when both control and intervention groups are given free antihypertensive medications and are involved in usual versus intensive intervention strategies. Because of this, it has not yet been determined whether the method of prescribing antihypertensive medications according to JNC 7 guidelines is more, less, or equally as effective as prescribing antihypertensive medications and providing intensive behavioral and clinical interventions. Knowledge in this area of HTN treatment should better able medical and health practitioners to help their AA subjects control HTN. The BEAT Hypertension Clinic will evaluate this method of HTN control by proposing a program that will evaluate the difference in HTN control among subjects receiving usual care and free medications and subjects also receiving free medications, but additionally being treated in a clinic that operates in a more intensive manner in relationship to patient behavior modification, patient-clinician interactions, and physical and social environments. At the conclusion of the study, the BEAT Hypertension Clinic investigators will report findings and help to answer the question of whether medication alone or medication combined with intensive behavioral and clinical treatment is more effective in HTN control in the AA population.

ELIGIBILITY:
Inclusion Criteria:

1. Demographics: men or women of self-declared African-American heritage between 25 and 80 years of age residing in the Omaha, Nebraska metropolitan area
2. History of documented uncontrolled (treated or untreated) hypertension (HTN) as defined by JNC 7 guidelines
3. Study eligibility will be based on the subject's current blood pressure control based on the average of two seated blood pressure measurements at two consecutive clinic visits at least one week apart

   1. Untreated subjects with elevated blood pressure (> 140/90 mmHg or < 130/80 mmHg for diabetics)
   2. Subjects treated with antihypertensive therapy whose blood pressure does not meet current JNC 7 guidelines (< 140/90 mmHg for non-diabetics and < 130/80 mmHg for diabetics)

Exclusion Criteria:

1. Myocardial infarction or stroke in the previous 6 months
2. Symptomatic heart failure or a left ventricular ejection fraction < 35%
3. Angina pectoris in the prior six months
4. Coronary revascularization procedure in the prior 6 months
5. Renal insufficiency defined as a serum creatinine > 2 mg/dl
6. Illicit drug or alcohol abuse in the prior 6 months
7. Dementia or other organic brain disease
8. Serious systemic illness with a shortened life expectancy or other limitation that precludes participation in this trial
9. Secondary HTN
10. Concurrent participation in an investigational medication trial

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2005-08; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syed Mohiuddin, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton Community Health Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 49 | 50
Completed | 49 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 47 | 93
  >=65 years | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 49.6 (9.81) | 50 (11) | 49.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 39 | 72
  Male | 16 | 11 | 27
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Blood Pressure Goals
Description: Percentage of subjects who achieved JNC-VII defined blood pressure goals.
Time Frame: 3 month intervals
Measure: Number; unit: percentage of participants
Groups:
- Intervention: Free antihypertensive medications, in-depth HTN and healthy living education, behavior change counseling, and Therapeutic Lifestyle Change following JNC-VII guidelines.
- Control: Free antihypertensive medications, basic hypertension education and usual clinical care.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 49 | 50
percentage of participants | 81 | 57

2. Secondary Outcome: New Onset Diabetes Mellitus
Time Frame: 3 month intervals
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes